CLINICAL TRIAL: NCT03091543
Title: A Double-blind, Randomised, Crossover, Placebo-controlled Study in Healthy Volunteers to Investigate the Tolerability, Safety and Pharmacokinetics of Four Single-doses of BIA 6-512 (Trans-resveratrol) and Their Effect on the Levodopa Pharmacokinetics When Administered in Combination With a Single-dose of Levodopa/Benserazide 100/25 mg
Brief Title: Tolerability, Safety and Pharmacokinetics of Four Single-doses of BIA 6-512 (Trans-resveratrol) and Their Effect on the Levodopa Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BIA-6512-101
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sequence A (25 mg - 50 mg - 100 mg - 200 mg - Placebo) (Experimental): Concomitantly with the BIA 6-512/Placebo dose, subjects will be administered levodopa/benserazide 100/25 mg. All subjects attended to each 5 treatment periods and received a different dose of BIA 6-512 or placebo in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg in each of these treatment periods. The washout period between periods was 5 days or more.
  Interventions: Drug: Madopar® HBS 125; Drug: Placebo; Drug: BIA 6-512 25 mg dose; Drug: BIA 6-512 50 mg dose; Drug: BIA 6-512 100 mg dose; Drug: BIA 6-512 200 mg dose
- Sequence B (Placebo - 25 mg - 50 mg - 100 mg - 200 mg) (Experimental): Concomitantly with the BIA 6-512/Placebo dose, subjects will be administered levodopa/benserazide 100/25 mg. All subjects attended to each 5 treatment periods and received a different dose of BIA 6-512 or placebo in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg in each of these treatment periods. The washout period between periods was 5 days or more.
  Interventions: Drug: Madopar® HBS 125; Drug: Placebo; Drug: BIA 6-512 25 mg dose; Drug: BIA 6-512 50 mg dose; Drug: BIA 6-512 100 mg dose; Drug: BIA 6-512 200 mg dose
- Sequence C (200 mg - Placebo - 25 mg - 50 mg - 100 mg) (Experimental): Concomitantly with the BIA 6-512/Placebo dose, subjects will be administered levodopa/benserazide 100/25 mg. All subjects attended to each 5 treatment periods and received a different dose of BIA 6-512 or placebo in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg in each of these treatment periods. The washout period between periods was 5 days or more.
  Interventions: Drug: Madopar® HBS 125; Drug: Placebo; Drug: BIA 6-512 25 mg dose; Drug: BIA 6-512 50 mg dose; Drug: BIA 6-512 100 mg dose; Drug: BIA 6-512 200 mg dose
- Sequence D (100 mg - 200 mg - Placebo - 25 mg - 50 mg) (Experimental): Concomitantly with the BIA 6-512/Placebo dose, subjects will be administered levodopa/benserazide 100/25 mg. All subjects attended to each 5 treatment periods and received a different dose of BIA 6-512 or placebo in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg in each of these treatment periods. The washout period between periods was 5 days or more.
  Interventions: Drug: Madopar® HBS 125; Drug: Placebo; Drug: BIA 6-512 25 mg dose; Drug: BIA 6-512 50 mg dose; Drug: BIA 6-512 100 mg dose; Drug: BIA 6-512 200 mg dose
- Sequence E (50 mg - 100 mg - 200 mg - Placebo - 25 mg) (Experimental): Concomitantly with the BIA 6-512/Placebo dose, subjects will be administered levodopa/benserazide 100/25 mg. All subjects attended to each 5 treatment periods and received a different dose of BIA 6-512 or placebo in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg in each of these treatment periods. The washout period between periods was 5 days or more.
  Interventions: Drug: Madopar® HBS 125; Drug: Placebo; Drug: BIA 6-512 25 mg dose; Drug: BIA 6-512 50 mg dose; Drug: BIA 6-512 100 mg dose; Drug: BIA 6-512 200 mg dose

INTERVENTIONS:
Drug: Madopar® HBS 125 — 1 capsule of Madopar® HBS 125 (levodopa 100 mg / benserazide 25 mg) in an open label manner, concomitantly with BIA 6-512/Placebo.
Drug: Placebo — 2 capsules of placebo
Drug: BIA 6-512 25 mg dose — 1 capsule of 25 mg plus 1 capsule of placebo
Drug: BIA 6-512 50 mg dose — 2 capsules of 25 mg
Drug: BIA 6-512 100 mg dose — 1 capsule of 100 mg plus 1 capsule of placebo
Drug: BIA 6-512 200 mg dose — 2 capsules of 100 mg

SUMMARY:
To investigate the effect of four single oral doses of BIA 6-512 (25 mg, 50 mg, 100 mg and 200 mg) on levodopa pharmacokinetics when administered in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg and to assess the tolerability and safety of four single oral doses of BIA 6-512 (25 mg, 50 mg, 100 mg and 200 mg) when administered in combination with a single-dose of controlled release levodopa/benserazide 100/25 mg.

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled, crossover study with five single-dose treatment periods, with a washout period between doses of 5 days or more. In each of the five consecutive treatment periods, eligible subjects were admitted to the UFH in the day prior to receiving the study medication. On the morning of the dosing day, subjects received BIA 6-512/Placebo concomitantly with Madopar® HBS 125 in fasting conditions (at least 8 hours) and remained in the UFH until at least 24 h post-dose; then, they were discharged and returned for the next period or the follow-up visit. Blood samples for the assay of plasma BIA 6-512, levodopa and 3-O-methyldopa (3-OMD) were taken at the following times: pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination (including neurological examination), and 12-lead ECG.
* Subjects who had clinical laboratory tests within normal reference values.
* Subjects who were negative for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who had negative for alcohol and drugs of abuse at screening and each admission to each treatment period.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, OR
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or first admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used prescription or over-the-counter medication within 2 weeks of first admission.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 4 months of their first admission.
* Subjects who had donated and/or received any blood or blood products within the previous 4 months prior to screening.
* Subjects who were vegetarians, vegans and/or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05-04 (Actual); Primary Completion 2004-07-23 (Actual); Study Completion 2004-07-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) post-dose - Levodopa | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of Levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Time of occurrence of Cmax (tmax) - Levodopa | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of Levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t), calculated by the linear trapezoidal rule - Levodopa | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of Levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞), calculated from AUC0-t + (Clast/λz), where Clast is the last quantifiable concentration and λz the apparent terminal rate constant - Levodopa | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of Levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Apparent terminal half-life, calculated from ln 2/λz (t1/2) - Levodopa | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of Levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Maximum observed plasma drug concentration (Cmax) post-dose - BIA 6-512 | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512 following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Time of occurrence of Cmax (tmax) - BIA 6-512 | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512 following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t), calculated by the linear trapezoidal rule - BIA 6-512 | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512 following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞), calculated from AUC0-t + (Clast/λz), where Clast is the last quantifiable concentration and λz the apparent terminal rate constant - BIA 6-512 | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512 following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Apparent terminal half-life, calculated from ln 2/λz (t1/2) - BIA 6-512 | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512 following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) post-dose - 3-OMD | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of 3-O-methyldopa (3-OMD) following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Time of occurrence of Cmax (tmax) - 3-OMD | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of 3-O-methyldopa (3-OMD) following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t), calculated by the linear trapezoidal rule - 3-OMD | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of 3-O-methyldopa (3-OMD) following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞), calculated from AUC0-t + (Clast/λz), where Clast is the last quantifiable concentration and λz the apparent terminal rate constant - 3-OMD | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of 3-O-methyldopa (3-OMD) following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg
Apparent terminal half-life, calculated from ln 2/λz (t1/2) - 3-OMD | pre-dose, ¼, ½, 1, 1½, 2, 3, 4, 6, 9, 12, 16 and 24 hours post-dose.
  Pharmacokinetic parameters of 3-O-methyldopa (3-OMD) following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or BIA 6-512 25 mg, 50 mg, 100 mg and 200 mg

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH), S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided